CLINICAL TRIAL: NCT05768139
Title: First-in-Human Study of STX-478, a Mutant-Selective PI3Kα Inhibitor as Monotherapy and in Combination With Other Antineoplastic Agents in Participants With Advanced Solid Tumors
Brief Title: First-in-Human Study of STX-478 as Monotherapy and in Combination With Other Antineoplastic Agents in Participants With Advanced Solid Tumors
Acronym: PIKALO-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 27691; J6M-OX-JSGA (Other: Eli Lilly and Company); STX-478-101 (Other: Scorpion Therapeutics, Inc); 2023-000442-41 (EudraCT Number); 2023-504807-94-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-01; First posted 2023-03-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Solid Tumors, Adult
Keywords: Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; HER2-negative breast cancer; HR-positive breast cancer; Gynecologic cancer; Endometrial cancer; Ovarian cancer; Cervical cancer; Head and neck cancer; Head and neck squamous cell carcinoma; Fulvestrant; Antineoplastic Agents; PI3Kα; PI3K alpha; PI3Kα mutation; Alpelisib; STX-478; PI3Kα inhibitor; Estrogen Receptor Antagonists; Estrogen Antagonists; Hormone Receptor Antagonists; Hormone Antagonists; Hormones, Hormone Substitutes, and Hormone Antagonists; Physiological Effects of Drugs; Palbociclib; Ribociclib; PIK3CA; PIK3CA mutation; Aromatase inhibitor; Letrozole; Anastrozole; Exemestane; Imlunestrant; Inavolisib; Capivasertib
MeSH Terms: conditions — Breast Neoplasms; Neoplasms by Site; Neoplasms; Breast Diseases; Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hereditary Sensory and Autonomic Neuropathies | interventions — STX-478; Fulvestrant; ribociclib; palbociclib; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Masking Description: In Part 1, Part 2 B0 and B2, and Part 3 C0, D0, and E0, participants are assigned to intervention. In Part 2 B1 and Part 3 C1, D1, and E1, participants are randomized to doses
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Advanced Solid Tumors) (Experimental): * Cohort A0: Advanced Solid tumors expressing PI3Kα mutations
  * Cohort A1: HR+ breast cancer expressing PI3Kα mutations
  Interventions: Drug: STX-478
- Dose Expansion (Experimental): * Cohort A1: HR+/HER2- breast cancer expressing PI3Ka mutations
  * Cohort A2: Gynecologic cancers
  * Cohort A3: Head and Neck Squamous Cell Carcinoma
  * Cohorts A4/A5: Other solid tumors not included in Cohorts A1, A2, or A3 expressing PI3Kα mutations
  * Cohort A6: Endometrial cancer
  Interventions: Drug: STX-478
- Dose Selection/Expansion: Combination STX-478 + fulvestrant (Experimental): Cohort B: HR+/HER2- or HR+/HER2low breast cancer expressing PI3Kα mutations
  Interventions: Drug: STX-478; Drug: Fulvestrant
- Dose Selection/Expansion Combination (Experimental): STX-478 + Endocrine therapy + CDK4/6 inhibitor Cohort C/D/E: HR+/HER2- or HR+/HER2low breast cancer expressing PI3Ka mutations
  Interventions: Drug: STX-478; Drug: Fulvestrant; Drug: Ribociclib; Drug: Palbociclib; Drug: Letrozole; Drug: Anastrozole; Drug: Exemestane

INTERVENTIONS:
Drug: STX-478 — STX-478 is a mutant-selective PI3Kα inhibitor
  Other Names: LY4064809
Drug: Fulvestrant — Fulvestrant
  Other Names: Faslodex
  Arms: Dose Selection/Expansion Combination; Dose Selection/Expansion: Combination STX-478 + fulvestrant
Drug: Ribociclib — Ribociclib
  Other Names: Kisqali
  Arms: Dose Selection/Expansion Combination
Drug: Palbociclib — Palbociclib
  Other Names: Ibrance
  Arms: Dose Selection/Expansion Combination
Drug: Letrozole — Letrozole
  Other Names: Femara
  Arms: Dose Selection/Expansion Combination
Drug: Anastrozole — Anastrozole
  Other Names: Arimidex
  Arms: Dose Selection/Expansion Combination
Drug: Exemestane — Exemestane
  Other Names: Aromasin
  Arms: Dose Selection/Expansion Combination

SUMMARY:
Study STX-478-101 (LY4064809) is a multipart, open-label, phase 1/2 study evaluating the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of STX-478 (LY4064809) in participants with advanced solid tumors with P13Ka mutations.

Part 1 will evaluate STX-478 as monotherapy in participants with advanced solid tumors. Part 2 will evaluate STX-478 therapy as combination therapy with fulvestrant in participants with hormone receptor positive (HR+) breast cancer. Part 3 will evaluate STX-478 as combination therapy with endocrine therapy (aromatase inhibitors, fulvestrant or imlunestrant) and a CDK4/6 Inhibitor (either Ribociclib, Palbociclib or Abemaciclib) in participants with HR+ breast cancer.

Each study part will include a 28-day screening period, followed by treatment with STX-478 monotherapy or combination therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Has an advanced or refractory solid tumor malignancy that is metastatic or locally advanced and unresectable (as specified by Cohort)
* Has a new or recent tumor biopsy (collected at screening, if feasible) or will provide an adequate tissue sample prior to screening
* Has a tumor that harbors a documented PI3Kα mutation (cohort specific criterion for cohort-specific mutation types)
* Is ≥18 years of age at the time of signing the ICF
* Has an ECOG performance status score of 0 or 1 at screening
* Has adequate organ function as defined per protocol

Key Exclusion Criteria:

* Has history (within ≤2 years before screening) of a solid tumor or hematological malignancy that is histologically distinct from the cancers being studied
* Has symptomatic brain or spinal metastases
* Has an established diagnosis of uncontrolled diabetes mellitus (defined as HbA1c ≥8% and/or FBG ≥140 mg/dL [7.7 mmol/L] and/or requiring or required insulin).
* Has had prior treatment with PI3K/AKT/mTOR inhibitor(s), except in certain circumstances
* Has had treatment with any local or systemic antineoplastic therapy or investigational anticancer agent within 14 days or 4 half-lives, whichever is longer, prior to the initiation of study treatment up to a maximum washout period of 28 days. Endocrine therapy does not require a washout period if the patient is enrolling in a cohort with the same combination endocrine therapy.
* Has toxicities from previous anticancer therapies that have not resolved to baseline levels or CTCAE grade ≤1, with the exception of alopecia and peripheral neuropathy.
* Has had radiotherapy within 14 days before the initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience at least 1 Dose Limiting Toxicity (DLT) | First 28 days of treatment
Proportion of participants who experience at least 1 DLT during the first 28 days of treatment | First 28 days of treatment
Cmax of STX-478 | 12 months
AUC(0-inf) of STX-478 | 12 months
AUC(0-t) of STX-478 | 12 months
AUC(0-τ) of STX-478 | 12 months
Change from baseline in ctDNA levels | 12 months
Changes in circulating markers of glucose metabolism as assessed by changes in circulating glycosylated hemoglobin (HbA1c) | 12 months
Changes in circulating markers of glucose metabolism as assessed by circulating fasting plasma glucose | 12 months
Changes in circulating markers of glucose metabolism as assessed by circulating C-peptide | 12 months
Objective response rate (ORR) defined as the percentage of participants with partial response or complete response based on RECIST 1.1 | 12 months
Incidence of TEAEs/SAEs ≥ grade 2 | 12 months
Frequency of TEAEs according to CTCAE v5.0 criteria | 12 months
Change in ECOG performance status | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (67):
- United States (29):
  - Ellison Clinic at Saint John's, Los Angeles, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Florida Cancer Specialists ORLANDO/DDU, Lake Mary, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UH Cleveland Medical Center, Cleveland, Ohio
  - Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - USO-Virginia Cancer Specialists, PC, Fairfax, Virginia
- Belgium (2):
  - Institut Jules Bordet, Anderlecht
  - UZ Leuven, Leuven
- France (6):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine-Lacassagne, Nice
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsmedizin Mannheim, Mannheim
- Mater Misericordiae Hospital, Dublin, Ireland
- Italy (9):
  - Azienda Ospedaliera Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - Spedali Civili di Brescia, Brescia
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa
  - Ospedale Santa Maria delle Croci, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Japan (4):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kansai Medical University Hospital, Hirakata
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - Kyoto University Hospital, Kyoto
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Erasmus MC, Rotterdam
- Spain (12):
  - Hospital Quiron Barcelona, Barcelona
  - South Texas Accelerated Research Therapeutics (START) Barcelona- HM Nou Delfos, Barcelona
  - Instituto Oncologico Dr Rosell (IOR), Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital San Pedro, Logroño
  - MD Anderson Cancer Center, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Universitari Sant Joan de Reus, Reus
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No